CLINICAL TRIAL: NCT01951183
Title: A MULTI-CENTER, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, PARALLEL-GROUP, PHASE 2A STUDY TO ASSESS THE EFFICACY AND SAFETY OF ONCE-DAILY RO6811135 IN TYPE 2 DIABETIC PATIENTS INADEQUATELY CONTROLLED WITH METFORMIN
Brief Title: A Study of RO6811135 in Patients With Type 2 Diabetes Who Are Inadequately Controlled With Metformin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Cancelled due to Sponsor's decision
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP29013
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO6811135 (Experimental)
  Interventions: Drug: RO6811135

INTERVENTIONS:
Drug: Placebo — RO681135 placebo subcutaneously daily
  Arms: Placebo
Drug: RO6811135 — Subcutaneously daily
  Arms: RO6811135

SUMMARY:
This multi-center, randomized, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy, safety and tolerability of RO6811135 in Type 2 diabetic patients treated with a stable dose of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the age of 18 and 65
* Have been diagnosed with diabetes for at least 3 months and treated with a stable dose of metformin for at least 8 weeks
* Hemoglobin A1c between 7.2 and 10.5%
* Fasting plasma glucose less than 250 mg/dL
* C-peptide greater than 1.5 ng/mL
* Body mass index (BMI) between 27 and 44

Exclusion Criteria:

* Pregnant or lactating women
* Type 1 diabetes
* Had undergone weight loss surgery or weight loss procedure involving the gastrointestinal tract, such as gastric bypass, gastric stapling, or gastric banding
* Uncontrolled hypertension or other significant cardiovascular disease as determined by investigator
* Significant kidney or liver disease as determined by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | from baseline to Week 12

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose (FPG) | from baseline to Week 12
Pharmacokinetics: Area under the concentration-time curve (AUC) | 12 weeks
Safety: Incidence of adverse events | 19 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche